CLINICAL TRIAL: NCT06930703
Title: Treatment of Sickle Cell Pain and Inflammation With Cannabidiol (SPICe)
Brief Title: Cannabidiol in Sickle Cell Disease
Acronym: SPICE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Susanna Curtis, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: STUDY-24-00903; IN123001222 (Other Grant/Funding Number: American Society of Hematology)
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-04

CONDITIONS: Sickle Cell Disease
Keywords: chronic pain; epidiolex; cannabidiol
MeSH Terms: conditions — Anemia, Sickle Cell; Chronic Pain | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Twice daily cannabidiol given at 3 dose levels, 200mg, 400mg, and 600mg, for 4 weeks, with 1:1:1:1 allocation of placebo to 3 drug doses.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Twice daily matching placebo
  Interventions: Drug: Placebo
- Cannabidiol 200 mg (Active Comparator): Twice daily 200 mg cannabidiol
  Interventions: Drug: Cannabidiol
- Cannabidiol 400 mg (Active Comparator): Twice daily 400 mg cannabidiol
  Interventions: Drug: Cannabidiol
- Cannabidiol 600 mg (Active Comparator): Twice daily 600 mg cannabidiol
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — Cannabidiol (CBD) twice daily taken orally for 4-weeks
  Other Names: Epidiolex
  Arms: Cannabidiol 200 mg; Cannabidiol 400 mg; Cannabidiol 600 mg
Drug: Placebo — Placebo equivalent twice daily taken orally for 4-weeks
  Arms: Placebo

SUMMARY:
Randomized, placebo-controlled, double masked, dose finding study of twice daily cannabidiol given at 3 dose levels, 200mg, 400mg, and 600mg, compared to placebo for 4 weeks.

DETAILED DESCRIPTION:
The researchers will conduct a randomized, double blind, placebo-controlled, study of cannabidiol in an oral formulation. Participants will be enrolled when they are not in pain crisis and have demonstrated a urine toxicology test free from cannabinoids in the past 30 days. The sample size will be 52 participants, aged ≥18, with 1:1:1:1 allocation of placebo to 3 drug doses. This is a dose finding study with a primary outcome of reduction of inflammatory cytokine TNFα.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Clinical diagnosis of SCD (HbSS, HbSC, HbSβ+; Thal, HbSβ0Thal, HbS variants)
* Baseline score of 60 or lower on the ASCQ-Me 7-day pain interference domain
* If on a SCD modifying therapy (hydroxyurea, regular blood transfusions, L-glutamine, voxelotor, crizanlizumab), on stable dose for at least 3 months
* If using opioids for pain at home, on stable dose for at least 3 months
* One urine toxicology negative for cannabinoids within 30 days of randomization
* Willing to abstain from cannabis, medical and illicit, during study weeks 1 through 4 • Not pregnant or nursing
* If a woman capable of becoming pregnant, willing to use a medically accepted form of birth control for the duration of study participation. Accepted forms include oral contraception, medroxyprogesterone, contraceptive implants or patch, surgical sterilization, total abstinence.
* Able to consent for research

Exclusion Criteria:

* No known intolerance to cannabinoids
* No history of psychotic episode, psychosis, or active suicidality
* No contraindication to epidiolex with attention to potential side effects, concurrent medications/substances, and concurrent medical problems, as evaluated by a physician
* Not a daily cannabis user
* No diagnosis of active substance use disorder
* No ALT>3 times the upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Tumor Necrosis Factor-alpha level | at 4 weeks
  Plasma levels of tumor necrosis factor-alpha, a marker of inflammation in sickle cell disease will be collected.

SECONDARY OUTCOMES:
Levels of Markers of Inflammation | at 4 weeks
  Levels of inflammatory markers (IL1a, IL1b, IL6, IL4 and IL10) will be collected.
White Blood Cell with differential | at 4 weeks
  The blood differential test measures the percentage of each type of white blood cell (WBC) that are in the blood. This test is done to diagnose an infection, anemia, or leukemia. It may also be used to monitor a condition or to see if treatment is working.
C-reactive protein level | at 4 weeks
  C-reactive protein (CRP) is produced by the liver. The CRP test is a general test to check for inflammation in the body. It is not a specific test. This means it can reveal that inflammation is present somewhere in the body, but it cannot pinpoint the exact location or reason.
Tryptase levels | at 4 weeks
  Tryptase is enzyme released by mast cells in the body during allergic reactions and other immune responses. Elevated levels in the blood can indicate severe allergic reactions (like anaphylaxis), mast cell disorders, or certain inflammatory conditions.
Substance P levels | at 4 weeks
  Substance P is neuropeptide that functions as a neurotransmitter and acts as a key mediator of pain sensation and inflammation in the body. It plays a role in various physiological processes including stress responses, mood regulation, and neurogenic inflammation.
Cytokines levels | at 4 weeks
  Cytokines is a protein measured in blood samples to assess the body's immune and inflammatory responses to treatment. Elevated or reduced levels can indicate how the immune system is reacting and may help determine treatment effectiveness or disease progression.
Adult Sickle Cell Quality of Life Measurement System | at 4 weeks
  The ASCQ-Me pain scale ranges from 0-100, with a standardized sickle cell disease population mean of 50 (standard deviation=10), where lower scores signify worse disease impact.
Patient Reported Outcome Information System (PROMIS) to measure Pain | at 4 weeks
  Patient Reported Outcome Information System (PROMIS) domains for pain impact, neuropathic pain, and nociceptive pain: A standardized patient-reported measure assessing different aspects of pain experience. The measure includes subscales for pain impact (0-40), neuropathic pain (0-30), and nociceptive pain (0-30), each evaluating distinct pain mechanisms and experiences. Total score ranges from 0-100, with higher scores indicating greater pain severity and impact on daily functioning. Results are reported as T-scores (population mean=50, standard deviation=10)
Leeds Assessment of Neuropathic Symptoms and Signs pain scale (S-LANSS) | 4 weeks
  Leeds assessment of neuropathic signs and symptoms
  The S-LANSS is a self-reported version of the Leeds Assessment of Neuropathic Symptoms and Signs pain scale. It aims to differentiate neuropathic pain (pain from nerve damage) from somatic or nociceptive pain (pain from body damage). Scores range from 0-24, with higher scores indicating greater pain.
Patient Reported Outcomes Measurement Information System (PROMIS) | at 4 weeks
  The PROMIS (Patient-Reported Outcomes Measurement Information System) for domains: Anxiety, Appetite, Nausea, and Cognitive function. The PROMIS measure is a brief, computer-adapted measure of symptoms for the domains. Each is a normalized measure with a mean of 50 and standard deviation of 10. Higher scores represent increased symptoms.
Oral Morphine Equivalents (OME) | at 4 weeks
  Oral Morphine Equivalents (OME)
Number of Emergency Room Visits | at 4 weeks
  Number of emergency room visits
Number of Hospital Admissions | at 4 weeks
  Number of hospital admissions
Number of Psychiatric Facility Utilizations | at 4 weeks
  Number of psychiatric facility utilization
Columbia-Suicide Severity Rating Scale - Severity and Intensity Subscale (C-SSRS SI) | at 4 weeks
  The C-SSRS rates an individual's degree of suicidal ideation (SI) on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The subscale identifies SI severity and intensity, which may be indicative of an individual's intent to commit suicide. C-SSRS SI ranges from 0 (no SI) to 5 (active SI with plan and intent). Higher score indicates more severity.
Prodromal Questionnaire - Brief Version (PQ-B) | at 4 weeks
  The Prodromal Questionnaire Brief Version (PQ-B) is a patient questionnaire that assesses the existence of a prodromal state or fully developed psychosis. The PQ-B includes 21 items that refer to thoughts, feelings and experiences that describe various symptoms, including abnormal perception, unconventional thinking, paranoia and negative symptoms. For each item, the participant is asked to indicate whether they had experienced that phenomenon in the past month (yes/no). The total score is calculated by summing the number of "yes" responses across all items. Full range is 0-21, with higher scores indicating a greater likelihood of experiencing prodromal symptoms or fully developed psychosis

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Curtis, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, Manhattan, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Specify Other Time FrameOn request.
Access Criteria: Researchers who provide a methodologically sound proposal. Any purpose. Proposals should be directed to Susanna.curtis@mssm.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link TBD).